CLINICAL TRIAL: NCT04209205
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group, Phase III Multicenter Study of Intravenous Secukinumab to Compare Efficacy at 16 Weeks With Placebo and to Assess Safety and Tolerability up to 52 Weeks in Subjects With Active Psoriatic Arthritis
Brief Title: Study to Demonstrate the Efficacy, Safety and Tolerability of Intravenous Secukinumab up to 52 Weeks in Subjects With Active Psoriatic Arthritis
Acronym: INVIGORATE 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIN457P12302
Record Dates: First submitted 2019-10-30; First posted 2019-12-24 (Actual); Results first posted 2024-04-26 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Psoriatic Arthritis
Keywords: Active Psoriatic Arthritis; Intravenous secukinumab; PsA
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This was a double-blind, randomized treatment trial.
  Subjects, investigator staff, persons performing the assessments remained blinded to the identity of the treatment from the time of randomization until Week 60 database lock, using the following methods:
  1. Randomization data were kept strictly confidential until the time of unblinding and were not accessible by anyone else involved in the study with the exception of the bioanalyst.
  2. The identity of the treatments were concealed by the use of study treatments in the form of i.v. injection, filled with secukinumab or placebo that were identical in appearance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AIN457 6 mg/kg - 3 mg/kg i.v. (Experimental): AIN457 6 mg/kg i.v. infusion at baseline, followed by AIN457 3 mg/kg i.v. infusion every 4 weeks starting at Week 4 through Week 48 (exposure through Week 52).
  Interventions: Drug: AIN457 6 mg/kg i.v.; Drug: AIN457 3 mg/kg
- Placebo (Placebo Comparator): Matching placebo from baseline to Week 16 and switch to AIN457 3mg/kg i.v. infusion every 4 weeks through Week 48 (exposure through Week 52).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AIN457 6 mg/kg i.v. — AIN457 6 mg/kg delivered by i.v. infusion
  Other Names: secukinumab
  Arms: AIN457 6 mg/kg - 3 mg/kg i.v.
Drug: Placebo — Matching placebo to AIN457 i.v. infusion
  Arms: Placebo
Drug: AIN457 3 mg/kg — AIN457 3 mg/kg delivered by i.v. infusion
  Other Names: secukinumab
  Arms: AIN457 6 mg/kg - 3 mg/kg i.v.

SUMMARY:
The purpose of this study was to provide up to 52 weeks of efficacy, safety and tolerability data to support registration of intravenous (i.v.) secukinumab (Initial dose of 6 mg/kg at Baseline (BSL) followed thereafter with 3 mg/kg administered every four weeks) in patients with active psoriatic arthritis (PsA) despite current or previous Non-steroidal anti-inflammatory drugs (NSAIDs), Disease-modifying antirheumatic drugs (DMARDs) and/or anti-tumor necrosis factor (TNF) therapy.

DETAILED DESCRIPTION:
This multicenter study used a randomized, double-blind, placebo-controlled, parallel-group design. A screening (SCR) period running up to 10 weeks before randomization was used to assess subject eligibility followed by a treatment period of 52 weeks.

At baseline, 381 patients with active psoriatic arthritis were randomized to one of the two treatment groups in a 1:1 randomization:

Group 1: Approximately 190 patients with active psoriatic arthritis; These patients received secukinumab 6 mg/kg i.v. at BSL, followed by the administration of secukinumab 3 mg/kg i.v. every four weeks starting at Week 4.

Group 2: Approximately 190 patients with active psoriatic arthritis; These patients received i.v. placebo at BSL and at Weeks 4, 8, and 12, followed by the administration of secukinumab 3 mg/kg i.v. every four weeks starting at Week 16.

Study consisted of 4 periods: a screening period (up to 10 weeks), treatment period 1 (total duration of 16 weeks) and treatment period 2 (total duration of 36 weeks) followed by a safety follow up period of 8 weeks after the end of treatment visit (i.e., Week 52).

Primary endpoint analysis will be performed with Week 16 data (last patient completing Treatment period 1 (Week 16). Long-term efficacy and safety assessments will be performed up to Week 52.

ELIGIBILITY:
Patients eligible for inclusion in this study had to fulfill all of the following criteria:

* Diagnosis of PsA classified by CASPAR criteria and with symptoms for at least 6 months with moderate to severe PsA who must have at Baseline ≥3 tender joints out of 78 and ≥3 swollen out of 76 (dactylitis of a digit counts as one joint each)
* Rheumatoid factor and anti-CCP antibodies negative at screening
* Diagnosis of active plaque psoriasis or nail changes consistent with psoriasis or documented history of plaque psoriasis
* Subjects with PsA should have taken NSAIDs for at least 4 weeks prior to randomization with inadequate control of symptoms or at least one dose if stopped due to intolerance to NSAIDs
* Subjects taking corticosteroids must be on a stable dose of ≤10 mg/day prednisone or equivalent for at least 2 weeks before randomization and should remain on a stable dose up to Week 16
* Subjects taking MTX (≤ 25 mg/week) are allowed to continue their medication if the dose is stable for at least 4 weeks before randomization and should remain on a stable dose up to Week 52.

Patients fulfilling any of the following criteria are not eligible for inclusion in this study:

* Chest X-ray or chest MRI with evidence of ongoing infectious or malignant process, obtained within 3 months prior to screening and evaluated by a qualified physician
* Subjects taking high potency opioid analgesics (e.g. methadone, hydromorphone, morphine)
* Previous exposure to secukinumab or other biologic drug directly targeting IL-17 or IL-17 receptor
* Ongoing use of prohibited psoriasis treatments / medications (e.g., topical corticosteroids, UV therapy) at randomization. The following wash-out periods need to be observed:
* Oral or topical retinoids- 4 weeks
* Photochemotherapy (e.g. PUVA)- 4 weeks
* Phototherapy (UVA or UVB)- 2 weeks
* Topical skin treatments (except in face, eyes, scalp and genital area during screening, only corticosteroids with mild to moderate potency)- 2 weeks
* Any intramuscular or intravenous corticosteroid treatment within 4 weeks before randomization.
* Any therapy by intra-articular injections (e.g. corticosteroid) within 4 weeks before randomization.
* Subjects who have previously been treated with more than 3 different TNF inhibitors (investigational or approved).
* Subjects who have ever received biologic immunomodulating agents, investigational or approved except for those targeting TNFα.
* Previous treatment with any cell-depleting therapies including but not limited to anti-CD20 or investigational agents (e.g., CAMPATH, anti-CD4, anti-CD5, anti-CD3, anti-CD19)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 381 (Actual)
Dates: Start 2020-01-29 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2022-05-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (74):
- United States (31):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Fountain Valley, California
  - Novartis Investigative Site, Fullerton, California
  - Novartis Investigative Site, La Mesa, California
  - Novartis Investigative Site, Santa Monica, California
  - Novartis Investigative Site, Upland, California
  - Novartis Investigative Site, Van Nuys, California
  - Novartis Investigative Site, West Hills, California
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Clearwater, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Ocoee, Florida
  - Novartis Investigative Site, Plantation, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Winter Park, Florida
  - Novartis Investigative Site, Marietta, Georgia
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Bowling Green, Kentucky
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Lincoln, Nebraska
  - Novartis Investigative Site, Voorhees Township, New Jersey
  - Novartis Investigative Site, Rochester, New York
  - Novartis Investigative Site, Greensboro, North Carolina
  - Novartis Investigative Site, Middleburg Heights, Ohio
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Tulsa, Oklahoma
  - Novartis Investigative Site, Duncansville, Pennsylvania
  - Novartis Investigative Site, Jackson, Tennessee
  - Novartis Investigative Site, Austin, Texas
  - Novartis Investigative Site, Mesquite, Texas
  - Novartis Investigative Site, Newport News, Virginia
- Brazil (2):
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, São Paulo, São Paulo
- Bulgaria (3):
  - Novartis Investigative Site, Burgas
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Sofia
- Colombia (4):
  - Novartis Investigative Site, Barranquilla, Atlántico
  - Novartis Investigative Site, Bucaramanga, Santander Department
  - Novartis Investigative Site, Bogotá
  - Novartis Investigative Site, Cundinamarca
- Czechia (2):
  - Novartis Investigative Site, Prague
  - Novartis Investigative Site, Uherské Hradiště
- Greece (2):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Thessaloniki
- Novartis Investigative Site, Guatemala City, Guatemala
- India (4):
  - Novartis Investigative Site, Surat, Gujarat
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Nashik, Maharashtra
  - Novartis Investigative Site, New Delhi
- Malaysia (3):
  - Novartis Investigative Site, Seremban, Negeri Sembilan
  - Novartis Investigative Site, Kuching, Sarawak
  - Novartis Investigative Site, Selangor Darul Ehsan
- Philippines (4):
  - Novartis Investigative Site, Lipa City, Batangas
  - Novartis Investigative Site, Dasmariñas, Cavite
  - Novartis Investigative Site, Manila
  - Novartis Investigative Site, Quezon City
- Poland (5):
  - Novartis Investigative Site, Krakow, Lesser Poland Voivodeship
  - Novartis Investigative Site, Karwiany
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Sochaczew
  - Novartis Investigative Site, Warsaw
- Russia (6):
  - Novartis Investigative Site, Kemerovo
  - Novartis Investigative Site, Nizhny Novgorod
  - Novartis Investigative Site, Rostov-on-Don
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Yaroslavl
  - Novartis Investigative Site, Yekaterinburg
- South Africa (2):
  - Novartis Investigative Site, Panorama, Western Cape
  - Novartis Investigative Site, Stellenbosch
- Thailand (4):
  - Novartis Investigative Site, Bangkoknoi, Bangkok
  - Novartis Investigative Site, Songkhla, Hat Yai
  - Novartis Investigative Site, Khon Kaen, THA
  - Novartis Investigative Site, Bangkok
- Novartis Investigative Site, Bursa, Gorukle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1500

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 479 participants were screened and and 381 were randomized.
Groups:
- Placebo to AIN457 3 mg/kg i.v.: Matching placebo from baseline to Week 16 and switch to AIN457 3 mg/kg i.v. infusion every 4 weeks through Week 48 (exposure through Week 52).
Period: Overall Study
Arm/Group | AIN457 6 mg/kg - 3 mg/kg i.v. | Placebo to AIN457 3 mg/kg i.v.
Started | 191 | 190
Completed | 173 | 167
Not Completed | 18 | 23
Not completed — Adverse Event | 2 | 3
Not completed — Lost to Follow-up | 3 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Subject decision | 10 | 10
Not completed — Progressive disease | 1 | 0
Not completed — Protocol deviation | 0 | 1
Not completed — New therapy for study indication | 1 | 0
Not completed — Adverse event - placebo not switched | 0 | 1
Not completed — Subject decision - placebo not switched | 0 | 5
Not completed — Death - placebo not switched | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomized set
Groups:
- Total: Total of all reporting groups
Arm/Group | AIN457 6 mg/kg - 3 mg/kg i.v. | Placebo to AIN457 3 mg/kg i.v. | Total
Number analyzed (Participants) | 191 | 190 | 381
Age, Customized [Number; unit: Participants]
  <65 years | 170 | 165 | 335
  65-74 years | 17 | 24 | 41
  >= 75 years | 4 | 1 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 105 | 209
  Male | 87 | 85 | 172
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 148 | 153 | 301
  Black or African American | 5 | 1 | 6
  Asian | 25 | 26 | 51
  American Indian or Alaska Native | 10 | 9 | 19
  More than one race | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With American College of Rheumatology 50 (ACR50) Response Comparison Between Treatment Groups Using Non-responder Imputation at Week 16 (Full Analysis Set)
Description: Percentage of participants with active psoriatic arthritis (PsA) who achieved an American College of Rheumatology 50 (ACR50) response
  The ACR50 is a composite measure defined as both improvement of 50% in the number of tender and number of swollen joints, and a 50% improvement in three of the following five criteria: patient global assessment, physician global assessment, functional ability measure [most often Health Assessment Questionnaire (HAQ)], visual analog pain scale, and erythrocyte sedimentation rate or C-reactive protein (CRP)
Time Frame: Baseline up to Week 16
Population: Full analysis set from which subset of ACR50 responders was analyzed
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | AIN457 6 mg/kg - 3 mg/kg i.v. | Placebo to AIN457 3 mg/kg i.v.
Number analyzed (Participants) | 191 | 190
Percentage of participants | 31.35 [24.80 to 37.90] | 6.33 [2.87 to 9.79]
Statistical Analysis 1: Comparison: AIN457 6 mg/kg - 3 mg/kg i.v. vs Placebo to AIN457 3 mg/kg i.v; Test type: Superiority; p < .0001, Regression, Logistic; Marginal difference = 25.02, 95% CI 2-sided [17.61 to 32.43]

2. Secondary Outcome: Percentage of Participants With American College of Rheumatology 20 (ACR20) Response Comparison Between Treatment Groups Using On-responder Imputation at Week 16 (Full Analysis Set)
Description: Percentage of participants with an American College of Rheumatology 20% (ACR20) response. A participant was a responder if the following 3 criteria for improvement from Baseline were met: • ≥ 20% improvement in 78 tender joint count; • ≥ 20% improvement in 76 swollen joint count; and • ≥ 20% improvement in at least 3 of the 5 following parameters: ◦ Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]); ◦ Patient's global assessment of disease activity (measured on a 100 mm VAS); ◦ Physician's global assessment of disease activity (measured on a 100 mm VAS); ◦ Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index (HAQ-DI)); ◦ C-Reactive Protein.
Time Frame: Baseline up to Week 16
Population: Full analysis set from which subset of ACR20 responders was analyzed
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | AIN457 6 mg/kg - 3 mg/kg i.v. | Placebo to AIN457 3 mg/kg i.v.
Number analyzed (Participants) | 191 | 190
Percentage of participants | 59.60 [52.67 to 66.52] | 29.01 [22.57 to 35.44]
Statistical Analysis 1: Comparison: AIN457 6 mg/kg - 3 mg/kg i.v. vs Placebo to AIN457 3 mg/kg i.v; Test type: Superiority; p < .0001, Regression, Logistic; Marginal difference = 30.59, 95% CI 2-sided [21.14 to 40.05]

3. Secondary Outcome: Percentage of Participants With Minimal Disease Activity (MDA 5/7) Comparison Between Treatment Groups Using On-responder Imputation at Week 16 (Full Analysis Set)
Description: MDA is assessed as 5 of the 7 following: ≤ 1 tender and swollen joint; entheseal count, PASI ≤ 1 or BSA ≤3%, PsA ≤ 15 and disease activity ≤ 20 (VAS) and HAQ-DI© ≤ 0.5
Time Frame: Baseline up to Week 16
Population: Full analysis set from which subset of MDA 5/7 responders was analyzed
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | AIN457 6 mg/kg - 3 mg/kg i.v. | Placebo to AIN457 3 mg/kg i.v.
Number analyzed (Participants) | 191 | 190
Percentage of participants | 22.45 [16.57 to 28.33] | 5.28 [2.10 to 8.46]
Statistical Analysis 1: Comparison: AIN457 6 mg/kg - 3 mg/kg i.v. vs Placebo to AIN457 3 mg/kg i.v; Test type: Superiority; p < .0001, Regression, Logistic; Marginal difference = 17.17, 95% CI 2-sided [10.48 to 23.85]

4. Secondary Outcome: Percentage of Participants With Psoriasis Area and Severity Index 90 (PASi90) Score for Patients With a >= 3% Body Surface Area Psoriasis at Baseline Using On-responder Imputation at Week 16 (Full Analysis Set)
Description: Change from baseline of a 90% reduction in the PASI score for patients with a >= 3% body surface area psoriasis at baseline. Four body surface areas are evaluated (head, trunk and upper and lower limbs) for plaque, erythema, scaling and thickness. The degree of severity of each sign in each of the 4 body areas was assigned a score of 0 to 4. Scores ranged from 0 to 72 and higher scores represent worsening severity.
Time Frame: Baseline up to Week 16
Population: Full analysis set from which subset of PASi90 responders was analyzed
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | AIN457 6 mg/kg - 3 mg/kg i.v. | Placebo to AIN457 3 mg/kg i.v.
Number analyzed (Participants) | 49 | 7
Percentage of participants | 47.85 [38.15 to 57.54] | 6.46 [1.83 to 11.09]
Statistical Analysis 1: Comparison: AIN457 6 mg/kg - 3 mg/kg i.v. vs Placebo to AIN457 3 mg/kg i.v; Test type: Superiority; p < .0001, Regression, Logistic; Marginal difference = 41.39, 95% CI 2-sided [30.64 to 52.13]

5. Secondary Outcome: Psoriatic Arthritis Disease Activity Score (PASDAS) Change From Baseline Using Mixed Model Repeated Measures (MMRM) at Week 16 (Full Analysis Set)
Description: PASDAS is a composite measure developed to assess disease activity in Psoriatic arthritis. It is calculated by utilizing seven measures: Patient reported measures (excluding mental component) (SF-36-PCS), skin, peripheral joint counts (tender and swollen joint counts), dactylitis (LDI), enthesitis (LEI), acute phase response (CRP), and patient and physician global VAS scores. The typical score range is between 0 and 10. Smaller values on PASDAS indicate a better condition; a negative change from baseline indicates improvement.
Time Frame: Baseline up to Week 16
Population: Full analysis set with participants with valid measures at baseline and Week 16
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | AIN457 6 mg/kg - 3 mg/kg i.v. | Placebo to AIN457 3 mg/kg i.v.
Number analyzed (Participants) | 175 | 170
scores on a scale | -2.24 (0.103) | -1.11 (0.103)
Statistical Analysis 1: Comparison: AIN457 6 mg/kg - 3 mg/kg i.v. vs Placebo to AIN457 3 mg/kg i.v; Test type: Superiority; p < .0001, Mixed Models Analysis; Least squares mean = -1.13, 95% CI 2-sided [-1.38 to 0.87], Standard Error of Mean 0.129

6. Secondary Outcome: Health Assessment Questionnaire - Disability Index (HAQ-DI) Score Change From Baseline Using Mixed Model Repeated Measures (MMRM) at Week 16 (Full Analysis Set)
Description: The Health Assessment Questionnaire - Disability Index is a patient-reported questionnaire consisting of 20 questions referring to eight domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and usual activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task are summed and averaged to provide an overall score ranging from 0 to 3, where zero represents no disability and three very severe, high-dependency disability. Negative mean changes from Baseline in the overall score indicate improvement in functional ability.
Time Frame: Baseline up to Week 16
Population: Full analysis set with participants with valid measures at baseline and Week 16
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | AIN457 6 mg/kg - 3 mg/kg i.v. | Placebo to AIN457 3 mg/kg i.v.
Number analyzed (Participants) | 181 | 183
scores on a scale | -0.39 (0.035) | 0.15 (0.035)
Statistical Analysis 1: Comparison: AIN457 6 mg/kg - 3 mg/kg i.v. vs Placebo to AIN457 3 mg/kg i.v; Test type: Superiority; p < .0001, Mixed Models Analysis; Least squares mean = -0.24, 95% CI 2-sided [-0.32 to 0.15], Standard Error of Mean -0.043

7. Secondary Outcome: Short Form 36-Physical Component Summary (SF36-PCS) Score Change From Baseline Using Mixed Model Repeated Measures (MMRM) at Week 16 (Full Analysis Set)
Description: The SF-36 is used to measure health-related quality of life with acute and chronic conditions. It consists of eight subscales that can be scored individually: Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, and Mental Health. Range of scoring is 0 -100, with higher scores indicating better health status.
Time Frame: Baseline up to Week 16
Population: Full analysis set with participants with valid measures at baseline and Week 16
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | AIN457 6 mg/kg - 3 mg/kg i.v. | Placebo to AIN457 3 mg/kg i.v.
Number analyzed (Participants) | 181 | 182
scores on a scale | 6.47 (0.558) | 2.34 (0.550)
Statistical Analysis 1: Comparison: AIN457 6 mg/kg - 3 mg/kg i.v. vs Placebo to AIN457 3 mg/kg i.v; Test type: Superiority; p < .0001, Mixed Models Analysis; Least squares mean = 4.13, 95% CI 2-sided [2.80 to 5.46], Standard Error of Mean 0.676

8. Secondary Outcome: Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Score Change From Baseline Using Mixed Model Repeated Measures (MMRM) at Week 16 (Full Analysis Set)
Description: The FACIT-Fatigue is a 13 item questionnaire that assesses self-reported fatigue and its impact upon daily activities and function. Response scale ranges from 0-4 and the total score range is 0 - 52. Higher scores indicate better quality of life
Time Frame: Baseline up to Week 16
Population: Full analysis set with participants with valid measures at baseline and Week 16
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | AIN457 6 mg/kg - 3 mg/kg i.v. | Placebo to AIN457 3 mg/kg i.v.
Number analyzed (Participants) | 181 | 183
scores on a scale | 6.15 (0.759) | 3.30 (0.750)
Statistical Analysis 1: Comparison: AIN457 6 mg/kg - 3 mg/kg i.v. vs Placebo to AIN457 3 mg/kg i.v; Test type: Superiority; p = 0.0024, Mixed Models Analysis; Least squares mean = 2.85, 95% CI 2-sided [1.01 to 4.68], Standard Error of Mean 0.933

9. Secondary Outcome: Modified Nail Psoriasis Severity Index (mNAPSI) Score Change From Baseline Using Mixed Model Repeated Measures (MMRM) at Week 16 (Full Analysis Set)
Description: The mNAPSI is an instrument to assess psoriatic nail involvement. Three groups of features (onycholysis and oil-drop dyshromia, pitting and crumbling) were graded on a scale from 0 to 3 for a total subscale of 0 to 9. The next 4 abnormalities (leukonychia, splinter hemorrhages, hyperkeratosis and red spots in the lunula) were graded as absent (0) or present (1) for a total subscale of 0 to 4. The total score was from 0-13 where higher scores represent worse nail disease.
Time Frame: Baseline up to Week 16
Population: Full analysis set with participants with valid measures at baseline and Week 16
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | AIN457 6 mg/kg - 3 mg/kg i.v. | Placebo to AIN457 3 mg/kg i.v.
Number analyzed (Participants) | 124 | 118
scores on a scale | -9.25 (1.069) | -3.14 (1.084)
Statistical Analysis 1: Comparison: AIN457 6 mg/kg - 3 mg/kg i.v. vs Placebo to AIN457 3 mg/kg i.v; Test type: Superiority; p < .0001, Mixed Models Analysis; Least squares mean = -6.11, 95% CI 2-sided [-8.96 to -3.26], Standard Error of Mean 1.447

10. Secondary Outcome: Percentage of Participants With Complete Resolution of Dactylitis at Week 16 Using Non-responder Imputation (Dactylitis Subset)
Description: Dactylitis is characterized by swelling of the entire finger or toe. The Leeds Dactylitis Index (LDI) measures the ratio of the circumference of the affected (swollen) digit. The ratio of circumference is multiplied by a tenderness score, using a modification of LDI that is a binary score (1 for tender, 0 for non-tender). The LDI requires a finger circumference gauge or a dactylometer to measure digital circumference. Scores range from 0 - 20 and lower score indicates better outcome.
Time Frame: Baseline up to Week 16
Population: Dactylitis subset - participants with dactylitis at baseline
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | AIN457 6 mg/kg - 3 mg/kg i.v. | Placebo to AIN457 3 mg/kg i.v.
Number analyzed (Participants) | 81 | 71
Percentage of participants | 59.53 [48.96 to 70.11] | 32.05 [21.33 to 42.76]
Statistical Analysis 1: Comparison: AIN457 6 mg/kg - 3 mg/kg i.v. vs Placebo to AIN457 3 mg/kg i.v; Test type: Superiority; p = 0.0003, Regression, Logistic; Marginal difference = 27.49, 95% CI 2-sided [12.43 to 42.55]

11. Secondary Outcome: Percentage of Participants With Complete Resolution of Enthesitis at Week 16 Using Non-responder Imputation (Enthesitis Subset (LEI))
Description: Enthesitis is inflammation of the enthesis which is where a a tendon or ligament attaches to the bone. The Leeds enthesitis index (LEI) is a validated index that uses 6 sites for evaluation of enthesitis: lateral epicondyle humerus L + R, proximal achilles L + R and medial condyle femur L+R. If enthesitis is present at any of the 6 sites, the subject is counted as a subject with enthesitis.
Time Frame: Baseline up to Week 16
Population: Enthesitis subset - participants with enthesitis at baseline
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | AIN457 6 mg/kg - 3 mg/kg i.v. | Placebo to AIN457 3 mg/kg i.v.
Number analyzed (Participants) | 126 | 110
Percentage of participants | 55.52 [46.92 to 64.12] | 39.16 [30.14 to 48.19]
Statistical Analysis 1: Comparison: AIN457 6 mg/kg - 3 mg/kg i.v. vs Placebo to AIN457 3 mg/kg i.v; Test type: Superiority; p = 0.0102, Regression, Logistic; Marginal difference = 16.35, 95% CI 2-sided [3.88 to 28.82]

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment up to a maximum of 481 days which included an approximate follow up period of 8 weeks for AIN457 treatment group.
Description: Any subjects randomized to Placebo were counted under 'Placebo' before being switched to AIN457 and under 'Any AIN457' after being switched to AIN457. It was pre-specified in the Study Protocol to monitor/assess Adverse Events irrespective of AIN457 dose level.
Groups:
- AIN457 6 mg/kg - 3 mg/kg i.v: AIN457 6 mg/kg i.v. infusion at baseline, followed by AIN457 3 mg/kg i.v. infusion every 4 weeks starting at Week 4 through Week 48 (exposure through Week 52). Includes participants switched from placebo at Week 16.
- Placebo up to Week 16: Matching placebo from baseline to Week 16
Arm/Group | AIN457 6 mg/kg - 3 mg/kg i.v | Placebo up to Week 16
All-Cause Mortality (participants affected / at risk) | 0/374 | 1/190
Serious Adverse Events (participants affected / at risk) | 22/374 | 4/190
Other Adverse Events (participants affected / at risk) | 136/374 | 35/190
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 6 mg/kg - 3 mg/kg i.v (N=374) | Placebo up to Week 16 (N=190)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
COVID-19 (Infections and infestations) | 6 | 0
COVID-19 pneumonia (Infections and infestations) | 2 | 2
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Perirectal abscess (Infections and infestations) | 1 | 0
Peritonsillar abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Viral pharyngitis (Infections and infestations) | 1 | 0
Procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 6 mg/kg - 3 mg/kg i.v (N=374) | Placebo up to Week 16 (N=190)
Diarrhoea (Gastrointestinal disorders) | 9 | 2
Nausea (Gastrointestinal disorders) | 11 | 2
Bronchitis (Infections and infestations) | 8 | 0
COVID-19 (Infections and infestations) | 37 | 7
Nasopharyngitis (Infections and infestations) | 13 | 3
Pharyngitis (Infections and infestations) | 9 | 1
Upper respiratory tract infection (Infections and infestations) | 10 | 6
Urinary tract infection (Infections and infestations) | 17 | 1
Alanine aminotransferase increased (Investigations) | 12 | 4
Aspartate aminotransferase increased (Investigations) | 11 | 2
Gamma-glutamyltransferase increased (Investigations) | 8 | 1
SARS-CoV-2 test positive (Investigations) | 12 | 2
Weight increased (Investigations) | 10 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 | 3
Headache (Nervous system disorders) | 12 | 5
Hypertension (Vascular disorders) | 12 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-09-24): https://cdn.clinicaltrials.gov/large-docs/05/NCT04209205/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-03): https://cdn.clinicaltrials.gov/large-docs/05/NCT04209205/SAP_001.pdf